CLINICAL TRIAL: NCT06850766
Title: A Randomized, Multicentre Pilot Trial Evaluating the Feasibility and Efficacy of Dose Timing (Morning vs Evening) of Temozolomide in the Treatment of Glioblastoma
Brief Title: The Feasibility and Efficacy of Dose Timing (Morning vs Evening) of Temozolomide in the Treatment of Glioblastoma
Acronym: TMZ-CHRONO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: The Ottawa Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TMZ-CHRONO
Record Dates: First submitted 2025-02-05; First posted 2025-02-27 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: IDH-Wildtype Glioblastoma; Glioblastoma (GBM)
Keywords: temozolomide; chronotherapy; dose timing; cancer; oncology; glioblastoma; chemotherapy
MeSH Terms: conditions — Glioblastoma; Neoplasms

STUDY DESIGN:
Intervention Model Description: Pragmatic pilot/feasibility trial.
Masking Description: Participants and investigators will not be blinded to treatment arm allocations due to the lack of placebo pills for TMZ in this study. The study aims to answer clinical questions using a pragmatic clinical trial design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Morning administration of TMZ (Active Comparator): Participants were instructed to take the prescribed daily dose of temozolomide (TMZ) in the morning.
  Interventions: Other: Morning administration of TMZ
- Evening administration of TMZ (Active Comparator): Participants were instructed to take the prescribed daily dose of temozolomide (TMZ) in the evening.
  Interventions: Other: Evening administration of TMZ

INTERVENTIONS:
Other: Morning administration of TMZ — Administration of TMZ within 2 hours of waking
  Arms: Morning administration of TMZ
Other: Evening administration of TMZ — Administration of TMZ within 2 hours of bedtime
  Arms: Evening administration of TMZ

SUMMARY:
The body's biological functions follow a circadian rhythm, meaning that individual biological functions in the body change over a 24-hour cycle. There is evidence suggesting that the body and cancer cells may react differently to anti-cancer treatment based on the time of day they are exposed. In fact, researchers have already found that giving anti-cancer treatments at a particular time of the day works better in rectal and ovarian cancer. Temozolomide (TMZ) is a chemotherapy pill/capsule commonly given to patients with newly diagnosed glioblastoma after brain surgery and radiation treatment. However, there is no current standard for what time of day TMZ should be taken for the treatment of glioblastoma.

In the current study, participants are randomly placed in one of two groups: a morning group and an evening group. Based on this group placement, participants are instructed to either take their TMZ in the morning or in the evening and record the date and time they take their TMZ in a pill diary. Participants will wear a wrist actigraphy device for the first cycle of TMZ. The primary goal of the study is to understand if taking TMZ at a prescribed time of day (morning/evening) is feasible in adults with glioblastoma. This is a pilot trial, and the investigators hypothesize that it will be feasible for glioblastoma patients to take TMZ at the prescribed time of day. The secondary goals of this study are to evaluate participant recruitment, safety, health-related quality of life, biological timing of TMZ delivery, and changes in condition over time. This pilot study will help investigators plan for a larger, pragmatic randomized clinical trial in the future.

DETAILED DESCRIPTION:
TMZ-CHRONO is a randomized, multi-centre pilot trial evaluating the feasibility of chronotherapy (dose-timing) for temozolomide (TMZ) in IDH-wildtype glioblastoma (GBM).

The body's biological functions follow a circadian rhythm. Chronotherapy is the deliberate timing of medications to enhance therapeutic benefit and/or minimize toxicity, and can be achieved by dose-timing treatments. There is evidence suggesting that cancer cells may react differently to chemotherapy based on the time of day they are exposed. In fact, researchers have already found that giving anti-cancer treatments at a particular time of the day works better in rectal and ovarian cancer. TMZ is a standard of care treatment for GBM, however there is currently no consensus or guideline with respect to the optimal timing of adjuvant TMZ administration. The study team recently conducted systematic review on TMZ chronotherapy in the treatment of glioma. With emerging evidence that TMZ timing may be important, it is paramount to conduct a large pragmatic randomized study to assess this claim in GBM. The current study is a minimal risk pilot trial to inform the development of a larger, pragmatic randomized clinical trial in the future.

Prospective participants will be approached by their physician (or a member within the circle of care) during their routine clinic visit to begin the integrated verbal consent model process. The physician will explain that the patient is receiving standard of care treatment, with the only change being the timing of adjuvant TMZ (morning vs evening). The physician will then ask the patient for verbal consent to participate in this research study and document this consent in the patient's electronic medical record. Eligible and consenting patients will be randomized to one of two study arms (morning administration of TMZ, and evening administration of TMZ) in a 1:1 fashion using a permuted block design through the Ottawa Methods Centre. Randomization will be stratified by cancer centre [The Ottawa Hospital Cancer Centre (TOHCC) and the London Health Sciences Centre (LHSC); Canada]. The participants and investigators will not be blinded to treatment arm allocations. The participants will wear a wrist actigraphy device during the first cycle of TMZ.

The primary aim of the study is to understand if taking TMZ at a prescribed time of day (morning/evening) is feasible in adults with GBM. The secondary aims of the study are to evaluate participant recruitment, safety, health-related quality of life, biological timing of TMZ deliver, and changes in condition over time. Data is collected throughout the study at baseline, randomization, pre/post-TMZ cycles, and at 4-, 8-, 12-, 24-, and 48-weeks after baseline. The study team will continue to follow the participant conditions after TMZ completion for up to 5 years.

This pilot trial is the first and necessary step to assess the feasibility of randomized treatment allocation, rate of pill diary completion, and metrics surrounding participant accrual. This will help determine the number of recruitment sites and expected duration of accrual for a future pragmatic, randomized clinical trial on chronotherapy of TMZ in IDH-wildtype GBM.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Newly diagnosed IDH-wildtype glioblastoma
* Completed maximal safe brain tumor resection
* Completed post-operative brain RT
* Plan to proceed with up to 6 cycles of adjuvant TMZ within 8 weeks of completing post-operative RT
* Able and willing to provide oral informed consent

Exclusion Criteria:

* Unable or unwilling to complete study questionnaires
* Metastatic or incurable cancer other than IDH-wild type glioblastoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-05-08 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2031-05 (Estimated)

PRIMARY OUTCOMES:
Feasibility: adherence to TMZ dose timing protocol | Patients complete daily pill diaries on days 1-5 of a 28-day cycle for up to 6 cycles. It is expected that the first cycle will begin within 8 weeks of the last fraction (dose) of radiation. Adherence is calculated at Week 48.
  The primary outcome is feasibility for patients to receive temozolomide (TMZ) according to their assigned dose timing. Feasibility is measured by at least 80% adherence to the assigned TMZ dose timing. Adherence is calculated based on patient entries in a daily pill diary.

SECONDARY OUTCOMES:
Participant recruitment: proportion of patients providing consent to participate | The number of patients providing consent to participate will be collected during the recruitment period and the total number/proportion will be calculated upon completion of recruitment. The anticipated recruitment period length is one year.
  The number of patients who provided consent for study participation over the total number of patients approached and invited to participate in the clinical study
Participant recruitment: participant withdrawal rate and reasons | Withdrawal rate and reasons will be collected from enrollment to start of adjuvant TMZ
  Proportion of eligible patients who consented to the study, but subsequently withdrew from study prior to starting the first cycle of adjuvant temozolomide (TMZ)
Participant recruitment: rate of patient enrollment | The number of patients enrolled in the study will be collected during the recruitment period. The anticipated recruitment period is one year.
  The rate of patient enrollment is defined by the number of new study participants who were randomized per center (average number of patients per month)
Safety: rate of hospital admissions | The number of hospitalizations will be collected from the start of adjuvant TMZ until 6 weeks after the last TMZ cycle (28-day cycles for up to 6 cycles). The number of hospitalizations per participant will be calculated at Week 48.
  Rate of hospital admissions per patient defined as the number of discrete admissions to acute care facility.
Safety: number of TMZ cycles | The number of TMZ cycles will be calculated at Week 48, once all questionnaires and adjuvant treatment cycles are complete.
  The median number of cycles received per group
Safety: reasons for early discontinuation of adjuvant TMZ | The reasons for early discontinuation of adjuvant TMZ will be collected during the treatment period: post-cycle 1, post-cycle 2, post-cycle 3, post-cycle 4, post-cycle 5. Each TMZ cycle is 28 days.
  The reasons for early discontinuation of adjuvant TMZ, if applicable, will be collected as a safety outcome.
Safety: rate of TMZ delay | TMZ delay is collected during the treatment period: post-cycle 1, post-cycle 2, post-cycle 3, post-cycle 4, post-cycle 5. Each TMZ cycle is 28 days. The rate of TMZ delay is calculated at Week 48.
  The rate of TMZ delay due to not meeting treatment parameters will be collected as a safety outcome.
Health-related quality of life (HR-QoL): FACT-Br Version 4 | Baseline and 4-, 8-, 12-, 24-, and 48-weeks after baseline.
  HR-QoL will be measured according to the Functional Assessment of Cancer Therapy -- Brain (FACT-Br) version 4. The FACT-Br includes five subscales: physical well-being (score range 0-28), social/family well-being (score range 0-28), emotional well-being (score range 0-24), functional well-being (score range 0-28), and brain cancer subscale (score range 0-92). The FACT-Br total scores range from 0 to 200. Higher scores indicate better quality of life.
HR-QoL: Time to HR-QoL deterioration | FACT-Br is collected at baseline and 4-, 8-, 12-, 24-, and 48-weeks after baseline..
  Time to health-related quality of life deterioration based on the Functional Assessment of Cancer Therapy - Brain (FACT-Br Version 4) Trial Outcome Index. The FACT-Br Trial Outcome Index includes physical well-being, functional well-being and brain subscales. The scores range from 0 to 148 and higher score indicate better quality of life.
Treatment-related side effects | Modified FACT-Br GP1, GP2, and GP5 are collected within 1 month of each TMZ cycle (28-day cycle). Post-cycle 1, post-cycle 2, post-cycle 3, post-cycle 4, post-cycle 5, post-cycle 6.
  Treatment related side effects are measured with modified Functional Assessment of Cancer Therapy - Brain items: GP1 lack of energy, GP2 nausea, GP5 bother by side effects. Each of the individual items are scored from 0 to 4, where higher scores indicate worse outcome.
Change in Trial Outcome Index | Baseline to 12-weeks
  Functional Assessment of Cancer Therapy - Brain (FACT-Br Version 4) Trial Outcome Index includes physical well-being, functional well-being and brain subscales. The FACT-Br Trial Outcome Index scores range from 0 to 148 and higher score indicate better quality of life. This outcome measure is a change in scores.
Change in FACT-Br scores | FACT-Br is collected at baseline and 4-, 8-, 12-, 24-, and 48-weeks after baseline.
  Change in mean Functional Assessment of Cancer Therapy - Brain (FACT-Br Version 4) scores from baseline between treatment groups. The FACT-Br total scores range from 0 to 200 and higher scores indicate better quality of life. This outcome measure is a change in scores.
Time to first progression | Disease assessment occurs prior to each TMZ cycle. Each TMZ cycle is 28 days. There is a maximum of 6 cycles.
  Time to first progression is defined as the time from randomization to time of investigator-assessed disease progression.
Overall survival | Overall survival is determined at 5-years after baseline.
  Overall survival (OS) is defined as the time from randomization to time of death. Time of death is collected through chart review and physician communications. Longitudinal follow-up will continue after completion of treatment until time of death or 5 years post-randomization for collection of overall survival data.
Internal biological time of TMZ delivery | Post-Cycle 1. Each cycle is 28 days in length.
  Daily internal biological time of TMZ delivery will be calculated based on actigraphy data (wrist movements in proportional integral mode) and clock timing of TMZ administration as recorded in the pill diary and with the actigraphy event marker.
Wall clock time of TMZ administration | Post-Cycle 1. Each cycle is 28 days in length.
  Wall clock time of TMZ administration is determined by self-reported pill diary entries and the actigraphy event marker.

CONTACTS AND LOCATIONS:
Overall Officials: Terry Ng, MD, Principal Investigator — The Ottawa Hospital Cancer Centre
Locations (2):
- Canada (2):
  - London Health Sciences Centre, London, Ontario
  - The Ottawa Hospital Cancer Centre, Ottawa, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jia JL, Alshamsan B, Ng TL. Temozolomide Chronotherapy in Glioma: A Systematic Review. Curr Oncol. 2023 Feb 4;30(2):1893-1902. doi: 10.3390/curroncol30020147. PMID 36826108
- See also: The Rethinking Clinical Trials (REaCT) website — https://react.ohri.ca/